CLINICAL TRIAL: NCT01495364
Title: A Prospective Randomized Double Blind Placebo Controlled Phase II Trial of Intra-coronary Infusion of AMR-001, a Bone Marrow Derived Autologous CD34+ Selected Cell Product, in Patients With Acute Myocardial Infarction.
Brief Title: NBS10 (Also Known as AMR-001) Versus Placebo Post ST Segment Elevation Myocardial Infarction
Acronym: PreSERVE-AMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lisata Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2011-12-09; First posted 2011-12-20 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: ST Segment Elevation Myocardial Infarction
Keywords: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NBS10 (Experimental): active treatment - CD34+ cells
  Interventions: Biological: NBS10
- placebo (Placebo Comparator): matching placebo
  Interventions: Other: placebo

INTERVENTIONS:
Biological: NBS10 — dosage = 10 or more million CD34+ cells via intracoronary infusion
  Other Names: AMR-001
  Arms: NBS10
Other: placebo — matching placebo
  Arms: placebo

SUMMARY:
This study will assess the safety and efficacy of intracoronary artery administered autologous bone marrow derived stem cells in subjects post ST segment elevation myocardial infarction (STEMI). This will be assessed by evaluating and comparing the autologous stem cell treatment group to the control group in terms of the occurrence of AE's, SAE's and Major Adverse Cardiac Events (MACE), by the change in myocardial perfusion (RTSS) measured quantitatively by gated single photon emission computed tomography myocardial perfusion imaging (gated SPECT MPI), and other secondary endpoints such as LVEF measured by cardiac MRI in addition to other endpoints.

DETAILED DESCRIPTION:
Efficacy endpoint is at 6 months. Clinical endpoints and safety will be measured through 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Acute ST elevation myocardial infarction meeting ACC/AHA criteria, with symptoms of chest pain within 3 days of admission. Criteria include (ST elevation > 1mm in limb leads or 2 mm in two or more precordial leads, and increased levels of troponin, CPK MB or both).

   Chest pain syndrome can extend to more than 3 days prior to admission if its course is consistent with transient/intermittent ischemia rather than symptoms that are continuous suggesting ongoing infarction extending beyond 3 days.
3. Successful stent placement and reperfusion within 3 days of chest pain onset and with TIMI Flow score of 2 or 3 and infarct related artery (IRA) with <20% stenosis after revascularization.
4. Wall motion abnormality associated with the target lesion
5. NYHA heart failure class I, II or III.
6. Study entry LVEF <48% determined by CMR no sooner than 96 hours from stent placement.
7. Able to provide informed written consent and willing to participate in all required study follow-up assessments.
8. Subjects must have an INR ≤ 2.0 within 2 days of the bone marrow collection.
9. Subjects must have a Hgb ≥ 10 grams/dL, WBC ≥ 3500 cells/mm3, a platelet count ≥ 100,000 cells/mm3, serum creatinine ≤ 2.5, and total bilirubin ≤ 2.0 within 7 days of the bone marrow collection or by end of screening phase.
10. Expected survival of at least one year.
11. Females of child bearing potential agree to use birth control (barrier method accepted) for one month post bone marrow harvest.

EXCLUSION CRITERIA

1. Continuous/ongoing chest pain - unremitting and unresponsive to nitroglycerin or rest - persisting 4 or more days before stent placement. If the chest pain syndrome is transient and/or intermittent - even if it began more than 3 days prior to admission - the patient is not excluded.
2. Subjects in cardiogenic shock (systolic pressure < 80mm/Hg, on vasopressors, or intra-aortic counterpulsation) at the time of consenting. Subjects who recover from cardiogenic shock by the time of consenting are eligible.
3. Subjects unable to receive antiplatelet agents (e.g. aspirin, clopidogrel, ticlopidine, prasugrel, etc).
4. Subjects receiving warfarin who have an INR >2 or with major bleeding requiring active transfusion support.
5. Subjects who require continuous anticoagulation during the time when the bone marrow harvest is scheduled, as heparin must be discontinued for 4 hours prior to and 24 hours after bone marrow harvest procedure. (See Appendix VII.)
6. Subjects with severe cardiac valvular disease expected to undergo surgery within 1 year.
7. Subjects with known severe immunodeficiency states (AIDS).
8. Cirrhosis requiring active medical management.
9. Malignancy requiring active treatment (except basal cell skin cancer).
10. Subjects with documented active alcohol and /or other substance abuse.
11. Females of child bearing potential unless a pregnancy test is negative within 7 days of the mini-bone marrow harvest.
12. Re-occlusion of the IRA prior to the infusion procedure.
13. Planned revascularization intervention during the next 6 months (A second PCI can be performed if done prior to qualifying CMR at least 96 hours post primary PCI).
14. Participation in an ongoing investigational trial.
15. Active or suspected bacterial infection requiring systemic intravenous antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2011-12; Primary Completion 2014-06 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
To determine safety and efficacy of intracoronary infusion of NBS10. | primary outcome measured at 6 months
  The primary endpoint includes the occurrence of AE's, SAE's and Major Adverse Cardiac Events (MACE) and the assessment of myocardial perfusion measured by quantitative gated SPECT MPI specifically looking at resting total severity score.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Moss, MD, Study Director — Lisata Therapeutics, Inc.; Arshed Quyyumi, MD, Principal Investigator — Emory University
Locations (58):
- United States (58):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Heart Center Research, LLC (Huntsville Hospital), Huntsville, Alabama
  - Mercy Gilbert Medical Group, Gilbert, Arizona
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - Scripps-La Jolla, CA, La Jolla, California
  - Keck School of Medicine - University of Southern California, Los Angeles, California
  - St.Johns Regional Hospital and Medical Center, Oxnard, California
  - Standford University School of Medicine, Stanford, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida-Gainesville, Gainesville, Florida
  - Orlando Health Medical Center, Orlando, Florida
  - Pepin Heart Institute - Florida Hospital -Tampa, Tampa, Florida
  - Emory University Medical Center, Atlanta, Georgia
  - St. Joseph's Research Institute, Atlanta, Georgia
  - Northeast Georgia Heart Center, Gainesville, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Advocate Health and Hospital Corp., Downer's Grove, Illinois
  - Advocate Health and Hospital Corp., Elmhurst, Illinois
  - St. Vincent's Medical Group/St. Vincent's Heart Center of Indiana, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Kentucky, Gill Heart Institute, Lexington, Kentucky
  - Louisville Cardiology Medical Group, Louisville, Kentucky
  - University of Maryland Med Center, Baltimore, Baltimore, Maryland
  - Metrowest Medical Center, Framingham, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Detroit Medical Center, Detroit, Michigan
  - Henry Ford Health Systems, Detroit, Michigan
  - Detroit Clinical Research Center PC, Farmington Hills, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Cardiology Asociates Research LLC, Tupelo, Mississippi
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Maimonides Medical Center-Brooklyn, Brooklyn, New York
  - Buffalo General Medical Center/Roswell Park Cancer Institute, Buffalo, New York
  - Stony Brook University Hospital and Medical Center, Stony Brook, New York
  - Westchester Medical Center, Valhalla, New York
  - Presbyterian CVI Research, Charlotte, North Carolina
  - CaroMont Heart, Gastonia, North Carolina
  - The Carl and Edyth Lindner Center for Research and Education at the Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Oklahoma Health and Sciences Center, Oaklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Drexel University/Hahnemann University Medical Center, Philadelphia, Pennsylvania
  - University of PIttsburg Medical Center, Pittsburgh, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - Stern Cardiovascular Foundation/Baptist Hospital, Memphis, Tennessee
  - Austin Heart, Austin, Texas
  - University of Texas Medical Branch - Galveston, Galveston, Texas
  - Texas Heart Institute, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Methodist Health Systems of San Antonio, San Antonio, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - UVA Health System Cardiology Research, Charlottesville, Virginia
  - Centra Lynchburg General Hospital, Lynchburg, Virginia
  - Aurora Health Care Metro, Inc/St. Lukes Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Quyyumi AA, Vasquez A, Kereiakes DJ, Klapholz M, Schaer GL, Abdel-Latif A, Frohwein S, Henry TD, Schatz RA, Dib N, Toma C, Davidson CJ, Barsness GW, Shavelle DM, Cohen M, Poole J, Moss T, Hyde P, Kanakaraj AM, Druker V, Chung A, Junge C, Preti RA, Smith RL, Mazzo DJ, Pecora A, Losordo DW. PreSERVE-AMI: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial of Intracoronary Administration of Autologous CD34+ Cells in Patients With Left Ventricular Dysfunction Post STEMI. Circ Res. 2017 Jan 20;120(2):324-331. doi: 10.1161/CIRCRESAHA.115.308165. Epub 2016 Nov 7. PMID 27821724